CLINICAL TRIAL: NCT03172845
Title: Prevalence of Vulnerable Plaque Its Location and Clinical Significance in Bifurcation Lesions Detected by Optical Coherence Tomography.
Brief Title: Optical Coherence Tomography (OCT) Findings and Coronary Bifurcation Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NFH20170423
Record Dates: First submitted 2017-05-11; First posted 2017-06-01 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Coronary Bifurcation Lesions
Keywords: coronary bifurcation lesion; optical coherence tomography; vulnerable plaque
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vulnerable plaque (Experimental): Thin-cap fibro atheroma (TCFA) was defined as a lipid-rich plaque with the thinnest fibrous cap thickness<65um. Plaque rupture was identified by the presence of fibrous cap discontinuity with a clear cavity formation inside the plaque. Plaque erosion is characterized by luminal thrombus and absence of the endothelium or without evidence of fibrous cap disruption. Fibro calcific plaque contains OCT evidence of fibrous tissue along with calcium that appears as a signal-poor or heterogeneous region with a sharply delineated border which is applied to larger calcifications. Calcified nodule is characterized as a signal or multiple regions of calcium protruding into the lumen, superficial calcification accompanied by substantive calcium proximal and or distal to the lesion. Thrombus is defined as a mass attached to luminal surface or floating within the lumen. It is seen as a protrusion inside the lumen of the artery with signal attenuation.
  Interventions: Procedure: percutaneous coronary intervention
- Without any vulnerable plaqueStable plaque (Active Comparator): patient with bifurcation lesion undergoing baseline coronary angiography and baseline OCT.
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — percutaneous coronary intervention with drug-eluting stent implantation.
  Other Names: PCI

SUMMARY:
To determine the clinical prevalence of vulnerable plaque using OCT in patients with coronary bifurcation lesion.

DETAILED DESCRIPTION:
This is a prospective registry study in which patient with bifurcation lesion undergoing baseline coronary angiography, baseline OCT and percutaneous coronary intervention will be studied. OCT is used to assess the prevalence of vulnerable plaque, its location at bifurcation lesions and compare vulnerable plaque related major adverse cardiovascular events (MACE) during one-year follow-up in bifurcation lesions between patients with vulnerable plaque and those without. Relationship between endothelial shear stress and vulnerable plaque. Relationship between bifurcation angle and vulnerable plaque.

Group A: presence of vulnerable plaque at the bifurcation Group B: absence of vulnerable plaque at the bifurcation Documentation of immediate post stent OCT and 12 months follow up angiography with OCT will be performed. Immediate post stent OCT to assess successful stent implantation and after 12 months follow up to document year major adverse cardiovascular events (MACE) included myocardial infraction, cardiac death and clinically driven target lesion revascularization, stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients with ischemic heart disease who are considered for coronary revascularization with PCI
* True coronary bifurcation lesion Medina 1.1.1, 0.1.1, 1.0.1 (stenosis> 50% by visual estimation) treated by drug-eluting stent
* Reference vessel diameter of main vessel >= 2.5mm and side branch >=2.0 mm by visual estimation

Exclusion Criteria:

* Saphenous vein grafts
* In-stent restenotic lesions
* Thombus-containing lesions
* Patient who had Myocardial infarction with in less than one month
* Patent who had bifurcation lesion dilation with balloon
* Contraindication or hypersensitivity to anti-platelet agents or contrast media
* Creatinine level ≥ 2.0 mg/dL
* Severe hepatic dysfunction (3 times normal reference values)
* Hemodynamic unstable patients
* Inability of OCT devise to cross the lesion into distal vessel
* Pregnant women or women with potential childbearing
* Inability to understand or read the informed content

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
The prevalence of coronary vulnerable plaques in bifurcation lesions using coherence tomography (OCT) | Documentation of baseline OCT
  Vulnerable plaque was considered when presence of Thin-cap fibro atheroma (TCFA), Lipid-rich plaque (vulnerable), Plaque rupture, Plaque erosion, thrombus and calcified nodule.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 0 to 12 months
  MACE was included myocardial infarction, cardiac death, and target lesion revascularization.
Stent Thrombosis | 0 to 12 months
  Stent thrombosis was defined according to the Academic Research Consortium definition.
Thin-cap fibroatheroma | 0 to 12 months
  Thin-cap fibroatheroma was defined as a lipid-rich plaque with the thinnest fibrous cap thickness < 65 µm.
Calcified nodule | 0 to 12 months
  Calcified nodule is characterized as a signal or multiple regions of calcium protruding into the lumen, superficial calcification accompanied by substantive calcium proximal and or distal to the lesion.
Plaque erosion | 0 to 12 months
  Plaque erosion is characterized by luminal thrombus and absence of the endothelium, without evidence of fibrous cap disruption.
Plaque rupture | 0 to 12 months
  Rupture was identified by the presence of fibrous cap discontinuity with a clear cavity formation inside the plaque.
Thrombus | 0 to 12 months
  Thrombus is defined as a mass attached to luminal surface or floating within the lumen. It is seen as a protrusion inside the lumen of the artery with signal attenuation.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, MD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No